CLINICAL TRIAL: NCT02519296
Title: A fMRI Study of the Treatment of Danish Veterans With Post-Traumatic Stress Disorder With Prolonged Exposure Therapy: Study Protocol for a Case-control Trial
Brief Title: A fMRI Study of the Treatment of Danish Veterans With PTSD With Prolonged Exposure Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Aagaard, MD, professor, senior consultant, DrMedSc, Aalborg University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE-PTSD-Klinik Syd
Record Dates: First submitted 2015-07-02; First posted 2015-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Observation; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolonged Exposure Therapy (Active Comparator): In total 30 Danish veterans will be recruited, who meet the ICD-10 diagnostic criteria for PTSD, and treated with PE.
  Intervention with eight sessions of PE, psychometrics, blood analyses and fMRI.
  Interventions: Behavioral: Prolonged Exposure Therapy; Behavioral: Observation; Device: fMRI
- 30 Danish veterans without PTSD (Active Comparator): A group of controls will be recruited consisting of age-appropriate same sex veterans who have participated in international missions similar to the patient group.
  Observation with psychometrics, blood analyses and fMRI.
  Interventions: Behavioral: Observation; Device: fMRI

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — 8 sessions with prolonged exposure therapy and fMRI.
  Arms: Prolonged Exposure Therapy
Behavioral: Observation — fMRI.
Device: fMRI — Functional Magnetic Resonance Imaging of the brain

SUMMARY:
In this article, the investigators report the design and protocol of a functional magnetic resonance imaging study (fMRI) of the treatment of Danish veterans with PTSD with Prolonged Exposure Therapy (PE). In total 30 Danish veterans will be recruited, who meet the ICD-10 diagnostic criteria for PTSD, and treated with PE. A group of controls will be recruited consisting of age-appropriate same sex veterans who have participated in international missions similar to the patient group

DETAILED DESCRIPTION:
Primary outcome measures are the changes in d2-test assessment of attention and concentration, Beck Depression Inventory, Post-traumatic Symptom Scale-Interview version and PTSD Checklist- Military Version.

Secondary outcome measures concern changes of Brain Derived Neurotrophic Factor (BNDF) and changes in the brain structure with focus on the hippocampal function using fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Danish veterans with ICD-10 diagnostic criteria for PTSD
* Controls: Danish veterans without ICD-10 diagnostic criteria for PTSD

Exclusion Criteria:

* Participants who have an active abuse of psychoactive substances with daily consumption.
* Participants who consume more than 21 units of alcohol per week, and who, during the last month, have had repetitive episodes with craving, episodes of loss of control due to alcohol consumption, and a weakened ability to manage consumption, stop or reduce consumption
* Participants who have a current ICD-10 diagnosis within:

  * F20 to F29 Schizophrenia
  * Schizotypical mental disorder
  * Delusional disorder
  * Acute and transient psychotic disorders and Schizoaffective psychosis
  * F30 Manic single episode
  * F31 Bipolar affective disorder
  * F60.2 Dyssocial personality structure
  * F60.3 Emotionally unstable personality structure
  * F90 Hyperkinetic disorder (ADHD) F98.8 Other behavioural and emotional disorders in childhood and adolescence (ADD)
* Participants who have a daily intake of sedative, anxiolytic
* Participants who score below 23 on the Mini Mental State Examination, and (5)
* Participants who within the last 3 months have had a serious suicide attempt.
* Exclusion criteria related to the fMRI scanning include:

  * Ferromagnetic prostheses (including straps prostheses, clips on blood vessels, pacemakers, and metal splinters)
  * claustrophobia and movements during the scan.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Psychometric changes | Baseline - 3-6-12-36 months
  Primary outcome measures are the changes in d2-test assessment of attention and concentration, Beck Depression Inventory, Post-traumatic Symptom Scale-Interview version and PTSD Checklist- Military Version.

SECONDARY OUTCOMES:
Biomedical changes | Baseline - end of treatment - 36 months
  Secondary outcome measures concern changes of Brain Derived Neurotrophic Factor (BNDF) and changes in the brain structure with focus on the hippocampal function using fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Kjølbye, MD, Study Chair — Aalborg University Hospital